CLINICAL TRIAL: NCT02936947
Title: Study to Evaluate the Benefit of a High Frequency Ventilation System During Lung or Breast Cancer Radiotherapy Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to Covid19 restrictions
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Jean Bourhis, Head of radio-oncology, Centre Hospitalier Universitaire Vaudois
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUV-DO-PART-2016
Record Dates: First submitted 2016-08-30; First posted 2016-10-18 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Lung Cancer; Breast Cancer
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tomotherapy (HFPV vs free breathing) (Experimental): Tomotherapy: locally advanced lung cancer (Stage III) or left breast cancer. High Frequency Percussive Ventilation will be coupled to tomotherapy treatment. The alternative procedure is free breathing.
  Interventions: Device: High Frequency Percussive Ventilation; Other: Free breathing
- linear accelerator (HFPV vs ABC) (Experimental): Linear accelerator: breast cancer or pulmonary cancers (Stage I/II) requiring a stereotaxic radiotherapy.
  High Frequency Percussive Ventilation will be coupled to linear accelerator. The alternative procedure is Active Breathing Control (ABC).
  Interventions: Device: High Frequency Percussive Ventilation; Other: Active Breathing Control

INTERVENTIONS:
Device: High Frequency Percussive Ventilation — High Frequency Percussive Ventilation
  Other Names: HFPV
Other: Free breathing — Free breathing
  Arms: tomotherapy (HFPV vs free breathing)
Other: Active Breathing Control — Active Breathing Control
  Other Names: ABC
  Arms: linear accelerator (HFPV vs ABC)

SUMMARY:
That study combines High Frequency Percussive Ventilation (HFPV) with radiotherapy treatment in patients with tumors that are moving with respiration like breast or lung cancers. The use of a High Frequency Percussive Ventilation system leads to the cessation of respiratory motions while administering radiotherapy (RT) to tumors which allows a reduction of the amount of irradiated normal tissues and which potentially decrease radiation-induced collateral damages.

DETAILED DESCRIPTION:
Primary objective :

Demonstrate the clinical benefit of the HFPV coupled to thoracic radiotherapy in 2 distinct and frequent clinical situations :

1. Tomotherapy for lung and left breast tumors. The investigators assume that the volume of irradiated healthy tissue will be much less when using HFPV as compared to free breathing during tomotherapy sessions .
2. In comparison with Active Breathing Control (ABC system). The investigators assume that the HFPV will lead to breathing motions cessation the same way as the ABC system, but will abrogate pause times when administrating the radiotherapy. This will shorten the radiotherapy sessions for lung patients treated with stereotaxis and for breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer eligible for tomotherapy or linear accelerator with ABC system
* lung cancer eligible for curative tomotherapy and with a significant breathing movements amplitude
* lung cancer eligible for ablative stereotaxis
* WHO 0 or 1

Exclusion Criteria:

* patients requiring oxygen or not able to lie on the back (dyspnea)
* pulmonary functions altered
* cardiac insufficiency
* patient not able to breathe with the High Frequency Ventilation System
* risk of pneumothorax when experiencing High Frequency Ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
HFPV vs free breathing: 1/3 decrease of V20 (lung) or 1/2 decrease of Dmax (breast) | 0-14 days between registration and treatment start according to standard patient care
  Radiotherapy treatment fractions (locally advanced lung: 33 fractions). Each patient will undergo a planning CT scan: one with HFPV and one without. The CT scan is done after the patient has been registered in the study and before treatment start.
  Dose distribution will be determined for both situations and patients will be treated with the most favourable one.
HFPV vs ABC: decrease the duration of radiotherapy fractions (lung: 1/2 and breast 1/3) | 0-14 days between registration and treatment start according to standard patient care
  Lung (5 fractions) or breast (25 fractions). Each patient will undergo a planning CT scan: one with HFPV and one without. The CT scan is done after the patient has been registered in the study and before treatment start.
  The time of fractions administration will be compared to theoretical times of treatment when patient is free breathing (lung 45 min for 12Gy/ breast 10 min for 2Gy).

CONTACTS AND LOCATIONS:
Overall Officials: Jean Bourhis, Prof, Principal Investigator — CHUV
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No